CLINICAL TRIAL: NCT00218244
Title: Treatment of Smokeless Tobacco Users: Use of Nicotine Replacement Products to Reduce Smokeless Tobacco Use
Brief Title: Using Smokeless Tobacco Products With Lower Nicotine Levels to Reduce Negative Effects of Smokeless Tobacco Use
Acronym: Brandswitch
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Dorothy Hatuskami, University of Minnesota
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIDA-14404-1; R01-14404-1; DPMC
Record Dates: First submitted 2005-09-16; First posted 2005-09-22 (Estimated); Last update posted 2017-01-10 (Estimated); Status verified 2008-06

CONDITIONS: Tobacco Use Disorder
Keywords: Brand Switching, smokeless tobacco use
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 Controlled use (Active Comparator): Reduction in tobacco toxicants by switching to a lower nicotine tobacco product under a controlled use condition.
  Interventions: Other: Lower Nicotine Smokeless Tobacco Product
- 2 Uncontrolled use (Active Comparator): Reduction in tobacco toxicants by switching to a lower nicotine tobacco product under an uncontrolled use condition.
  Interventions: Other: Lower Nicotine Smokeless Tobacco Product
- 3 Behavioral (Placebo Comparator): Reduction in smokeless tobacco use using behavioral techniques only.
  Interventions: Other: Behavioral Counseling

INTERVENTIONS:
Other: Lower Nicotine Smokeless Tobacco Product — Skoal for 50% reduction;Skoal bandits for 75% reduction.
  Other Names: Skoal and Skoal Bandits
  Arms: 1 Controlled use; 2 Uncontrolled use
Other: Behavioral Counseling — Behavioral counseling alone for reduction in tobacco use.
  Arms: 3 Behavioral

SUMMARY:
Though spit tobacco is smokeless, it still affects the cardiovascular system and may be associated with heart disease, stroke, and high blood pressure. This study will assess the effectiveness of limiting smokeless tobacco (ST) nicotine intake in reducing levels of exposure to tobacco and associated toxicity, as well as enhancing motivation to either quit or sustain lower levels of nicotine intake.

DETAILED DESCRIPTION:
Spit tobacco presents as many health risks to its users as smoking tobacco. It affects the cardiovascular system and may be associated with heart disease, stroke, and high blood pressure. Long-term effects of spit tobacco use include tooth abrasion, gum recession, mouth disease, bone loss in the jaw, yellowing of the teeth, and chronic bad breath. Although a significant number of ST users recognize the importance of quitting, many either do not want to quit or feel it is impossible. For these individuals, tobacco reduction may be an important transitional goal, either prior to quitting, or as a treatment endpoint; however, approaches to help ST users reach this goal have not been studied. This study will assess the effectiveness of limiting ST nicotine intake in reducing levels of exposure to tobacco and associated toxicity, as well as enhancing motivation to either quit or sustain lower levels of nicotine intake.

Participants in this open-label study will be randomly assigned to one of three treatment conditions: switching to an ST brand with less concentrated nicotine and controlling for ST use; switching to an ST brand with less concentrated nicotine, combined with no limit on ST intake; or continued use of usual ST brand with no limit on intake (control group). Participants in both brand-switching conditions will use ST brands that have 50% less nicotine than their usual ST brands for the first 4 weeks. For the next 4 weeks, participants in the brand-switching conditions will use ST brands that have 75% less nicotine that their usual ST brands. Study visits will ocur once weekly during the 8-week treatment period. The number of participants who do not complete treatment, reduce nicotine intake, or quit completely will be assessed at Week 8 and at follow-up visits, which will be held 12 and 26 weeks following the completion of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Not interested in quitting ST use within 90 days of study entry
* Has been using ST at least six times a day for 6 months prior to study entry
* Agrees to use an effective form of contraception throughout the study

Exclusion Criteria:

* Current use of other tobacco or nicotine products
* Pregnant or breastfeeding
* Any unstable medical condition
* Use of any medication that may affect tobacco use or be affected by reduction of tobacco use
* DSM-IV diagnosis of any psychiatric disorders or substance abuse disorders within 6 months prior to study entry
* Use of any psychotropic medications within 6 months prior to study entry

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2001-08; Primary Completion 2004-11 (Actual); Study Completion 2004-11 (Actual)

PRIMARY OUTCOMES:
Percent reduction in ST use | 26 weeks
Toxicity profile of carcinogen metabolites | 26 weeks
Number of unsuccessful quit attempts | 26 weeks
Abstinence from ST use (measured at Week 8, and 12 and 26 weeks following treatment completion) | 26 weeks

SECONDARY OUTCOMES:
Motivation and self-efficacy (measured at Week 8, and 12 and 26 weeks following treatment completion) | 26 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dorothy Hatsukami, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States